CLINICAL TRIAL: NCT04361344
Title: Neurodegeneration Markers and Neurological Course in Severe Covid-19 Infection - MARNEVO-Covid
Brief Title: Neurodegeneration Markers and Neurological Course in Severe Covid-19 Infection
Acronym: MARNEVO-Covid
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: objective of the study demonstrated by other research teams
Sponsor: Centre Hospitalier de PAU (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHPAU2020/02
Record Dates: First submitted 2020-04-16; First posted 2020-04-24 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: COVID-19 Infection; Encephalitis
Keywords: COVID-19; encephalitis; biomarkers; neurofilament protein light; GFAP protein
MeSH Terms: conditions — COVID-19; Encephalitis | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Prospective, descriptive, monocentric, non-controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: blood samples — Clinical examination and blood samples will be done at inclusion (day 0), at day 7 (between day 4 and exit from intensive care) and at day 60.

SUMMARY:
Emergence of Covid-19 virus is associated with high frequency of extremely severe clinical pictures, with minor signs of CNS impairment (e.g. anosmia, headache). Since neurotropism is a common feature of coronavirus infection in animals, the investigators examine if indirect signs of CNS lesion are observed in association with severe Covid-19 infection.

DETAILED DESCRIPTION:
In animals, coronavirus infection is commonly associated with CNS involvement:

epilepsy and ataxia are observed during Feline Infectious Peritonitis (FIP) and virus is recovered in CSF, CNS is involved with strain-dependent severity in mice and rats infected by murine hepatitis virus, and murine infection with MHV A59 strain is a model of multiple sclerosis (MS). Mice encephalitis occurs through infection of olfactory bulb and spreads along the axonal pathway. Viral antigens and neuronal apoptosis are observed in brainstem and hypothalamus, without minimal or absent inflammation.

Most COVID-19 patients with neurologic impairment displayed expected complications of severe infections (e.g. neuropathy and muscle loss, stroke) but encephalitis remained exceptional, as previously observed in SRAS. It is argued that central lesions may explain some of the clinical features ventilation failure, or disproportionate residual fatigue and cognition impairment in survivors of severe COVID infection. According to data obtained from various coronavirus infections in animals, the investigators ask if severe COVID infection in human could be associated with sub-clinical encephalitis. This clinical trial examines highly sensitive blood biomarkers of brain dysfunction in correlation with late clinical outcome. Biomarkers are neurofilament light chain (NFL) and GFAP. Clinical outcomes are death, signs of central neurologic sequellae, and fatigue. Clinical examination and blood samples will be obtained at inclusion (d0), which is mostly the entrance in intensive care unit (ICU), at day 7 (between day 4 and exit from ICU) and at day 60.

ELIGIBILITY:
Inclusion Criteria:

* Infection with Covid-19 (proven or probable) AND
* possible encephalitis (at least confusion, epilepsy) OR
* clinical severity requiring invasive ventilation.

Exclusion Criteria:

* brain stroke
* minor CNS dysfunction (isolated smell loss or headache),
* absence of Covid infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2020-10-25 (Actual); Study Completion 2020-10-25 (Actual)

PRIMARY OUTCOMES:
Change of neurodegeneration markers level | Level of neurofilament light chain (NFL) is dosed at inclusion (day 0) and week 1. Level of GFAP is dosed at inclusion (day 0) and week 1 (day 7).
  Change of neurofilament light chain (NFL) (pg/ml) level between first day of hospitalisation and one week; and change of GFAP (pg/ml) level between first day of hospitalisation and one week.

CONTACTS AND LOCATIONS:
Locations (1):
- CH de Pau, Pau, France